CLINICAL TRIAL: NCT03662789
Title: Intravenous Iron Supplement for Iron Deficiency in Cardiac Transplant Recipients
Acronym: IronIC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Pharmacosmos A/S (Industry)
Responsible Party: Principal Investigator, Lars Gullestad, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IronIC
Record Dates: First submitted 2018-04-17; First posted 2018-09-07 (Actual); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-04

CONDITIONS: Heart Transplant Recipients
Keywords: Heart transplant; Iron deficiency; Intravenous iron supplement; Peak oxygen consumption; Cardiopulmonary exercise test; Cognitive function; Muscle strength
MeSH Terms: conditions — Iron Deficiencies | interventions — iron isomaltoside 1000

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, parallel group, double blind design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Opaque envelopes, infusion administered by third party, concealed infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iron isomaltoside 1000 (Active Comparator): The active drug, iron isomaltoside 1000 will be administered as a single, intravenous infusion of 20 mg/kg body weight (rounded off to the nearest 100 mg) dissolved in 100 ml NaCl as recommended by the drug manufacturer ("on-label" treatment).
  Interventions: Drug: Iron Isomaltoside 1000
- Placebo (Placebo Comparator): Patients allocated to placebo will receive an intravenous infusion of 100 ml NaCl 0.9%
  Interventions: Other: Placebo: NaCl 0,9%

INTERVENTIONS:
Drug: Iron Isomaltoside 1000 — Intravenous infusion
  Other Names: Monofer B03AC-
  Arms: Iron isomaltoside 1000
Other: Placebo: NaCl 0,9% — Intravenous infusion
  Arms: Placebo

SUMMARY:
Iron deficiency is prevalent in heart transplant recipients, and may be associated with reduced functional capacity. The IronIC trial is designed to assess the effect of intravenous iron isomaltoside on exercise capacity, muscle strength, cognition and quality of life in iron-deficient heart transplant recipients

DETAILED DESCRIPTION:
Iron deficiency is prevalent in patients with heart failure. Iron deficiency is associated with a worse prognosis, and randomised controlled trials have shown that correction of iron deficiency with intravenous iron therapy improves functional capacity, quality of life, and 6-minute walk distance. Current guidelines therefore recommend intravenous iron substitution in patients with heart failure with reduced ejection fraction and iron deficiency. Intravenous iron is more effective, better tolerated, and improves quality of life to a greater extent than oral iron supplements. In the IRONOUT HF trial, in which 225 patients with systolic heart failure were randomised to oral iron supplement or placebo, there was no effect on oxygen uptake, 6-minute walk distance, or quality of life. The authors attributed the negative results to the minimal effect on iron stores, suggesting that oral iron does not adequately replenish iron stores in patients with heart failure.

Cardiac allograft recipients resemble patients with heart failure in many respects. Prior to transplantation, and in some instances after heart transplantation, they have had overt heart failure. Moreover, due to the immunologic challenge posed by the allograft, and their susceptibility to infection due to immunosuppressive treatment, cardiac allograft recipients have low-grade inflammation. This low-grade inflammation makes it difficult to interpret iron stores, and results in dysregulated iron metabolism.

There have been no studies to assess the effect of intravenous iron therapy in heart transplant recipients who have iron deficiency. There is reason to believe that a liberal definition of iron deficiency should be used in cardiac allograft recipients, and the investigators have elected to use the well-established definition used in patients with heart failure: serum ferritin < 100 µg/l or ferritin between 100 and 300 µg/l in combination with a transferrin saturation < 20 %. Because oral iron supplement is less effective then intravenous iron in general, and in patients with heart failure in particular, the investigators assume that oral iron supplement is inadequate in heart transplant recipients. the investigators have designed the IronIC trial to assess the effect of intravenous iron isomaltoside on exercise capacity, muscle strength, cognition and quality of life in iron-deficient heart transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac allograft.
* Presentation at least one year after heart transplantation.
* Iron deficiency defined as serum ferritin < 100 µg/l or ferritin between 100 and 300 µg/l in combination with a transferrin saturation < 20 %.
* Age between 18 and 80 years.
* Informed consent obtained and documented according to Good Clinical Practice (GCP), and national/regional regulations.

Exclusion Criteria:

* Anaemia (Haemoglobin < 100 mg/l)
* Haemochromatosis
* Haemosiderosis
* Porphyria cutanea tarda
* Blood dyscrasias or any disorders causing haemolysis or unstable red blood cells
* Decompensated liver disease (Child-Pugh score 7 or higher)
* End-stage renal failure, i.e. estimated glomerular filtration rate < 15 ml/min or on renal replacement therapy
* Planned cardiac surgery or angioplasty within 6 months
* Planned major surgery within 6 months
* Medical history of unresolved cancer (except for basal cell carcinoma)
* Treatment with systemic steroids more than the equivalent of 10 mg Prednisone/day at the time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent
* Any uncontrolled endocrine disorder except type 2 diabetes
* Pregnancy
* On erythropoietin analogues
* Known sensitivity or intolerance to iron isomaltoside or other parenteral iron preparations
* Intravenous iron supplement within 6 months prior to inclusion
* On oral iron substitution (unless the subject agrees to stop treatment prior to randomisation)
* Ongoing rejections or infections
* Alcohol or drug abuse within 3 months of informed consent that would interfere with trial participation or any ongoing condition leading to decreased compliance with study procedures or study drug intake
* Intake of an investigational drug in another trial within 30 days prior to intake of study medication in this trial or participating in another trial involving an investigational drug and/or follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Gullestad, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo university Hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brautaset Englund KV, Ostby CM, Rolid K, Gude E, Andreassen AK, Gullestad L, Broch K. Intravenous iron supplement for iron deficiency in cardiac transplant recipients (IronIC): A randomized clinical trial. J Heart Lung Transplant. 2021 May;40(5):359-367. doi: 10.1016/j.healun.2021.01.1390. Epub 2021 Jan 23. PMID 33612360
- [Derived] Burker BS, Brautaset Englund KV, Myrdal Ostby C, Andersson S, Gullestad L, Broch K. Cognitive Function Among Heart Transplant Recipients Before and After Intravenous Iron Supplement for Iron Deficiency: Results From a Randomized, Placebo-Controlled, Double-Blind Treatment Trial. Clin Transplant. 2025 Nov;39(11):e70370. doi: 10.1111/ctr.70370. PMID 41182019

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iron Isomaltoside 1000 | Placebo
Started | 52 (Baseline) | 50 (Baseline)
Completed | 47 (Follow-up at 6 months) | 43 (Follow-up at 6 months)
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 1 | 2
Not completed — Could not perform treadmill test | 4 | 4
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Isomaltoside 1000 | Placebo | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 39 | 73
  >=65 years | 18 | 11 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (15) | 55 (14) | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 34 | 31 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 52 | 50 | 102
Peak oxygen consumption [Mean (Standard Deviation); unit: ml/kg/min] | 24.3 (7.3) | 22.3 (6.0) | 23.4 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Peak Oxygen Consumption
Description: The primary endpoint will be the baseline-adjusted between-group difference in peak oxygen consumption as measured on a treadmill exercise test
Time Frame: 6 months after intervention
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Iron Isomaltoside 1000 | Placebo
Number analyzed (Participants) | 47 | 43
ml/kg/min | 23.9 (6.6) | 22.0 (6.1)

2. Secondary Outcome: Iron Deficiency
Description: The number of patients with absolute or functional iron deficiency
Time Frame: 6 months after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside 1000 | Placebo
Number analyzed (Participants) | 47 | 43
Participants | 7 | 40

3. Secondary Outcome: Muscle Strength
Description: Baseline-adjusted muscle strength as measured by a hand-grip dynamometer
Time Frame: 6 months after intervention
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Iron Isomaltoside 1000 | Placebo
Number analyzed (Participants) | 47 | 43
kg | 40 (13) | 38 (12)

4. Secondary Outcome: Health Related Quality of Life: SF-36, Physical Component Summary (PCS)
Description: Baseline-adjusted quality of life as assessed with the 36-item short form survey (SF-36), which measures each of the following 8 health domains: 1= general health, 2= physical function, 3= role physical, 4= bodily pain, 5= vitality, 6= social function, 7= role emotional, 8= mental health. Total score for each domain are scaled 0 (minimum) to 100 (maximum), where higher scores represented higher level of functioning. Two norm-based sum scores, the physical and the mental component summaries with a mean of 50±10, were generated from the eight scale scores using a T-score transformation. Higher scores represented higher level of functioning.
Time Frame: 6 months after intervention
Measure: Median (Inter-Quartile Range); unit: t-score
Arm/Group | Iron Isomaltoside 1000 | Placebo
Number analyzed (Participants) | 47 | 43
t-score | 49 [42 to 55] | 45 [37 to 53]

5. Secondary Outcome: N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP)
Description: The between-group difference in baseline-adjusted NT-proBNP
Time Frame: 6 months after intervention
Measure: Median (Inter-Quartile Range); unit: ng/l
Arm/Group | Iron Isomaltoside 1000 | Placebo
Number analyzed (Participants) | 47 | 43
ng/l | 421 [134 to 807] | 349 [237 to 706]

6. Secondary Outcome: Cardiac Troponin T (TnT)
Description: The between-group difference in baseline-adjusted TnT
Time Frame: 6 months after intervention
Measure: Median (Inter-Quartile Range); unit: ng/l
Arm/Group | Iron Isomaltoside 1000 | Placebo
Number analyzed (Participants) | 47 | 43
ng/l | 13.0 [8.0 to 25.8] | 15.0 [8.0 to 24.3]

7. Secondary Outcome: Health Related Quality of Life: SF-36, Mental Component Summary (MCS)
Description: as for outcome 4
Time Frame: 6 months after intervention
Measure: Median (Inter-Quartile Range); unit: t-score
Arm/Group | Iron Isomaltoside 1000 | Placebo
Number analyzed (Participants) | 47 | 43
t-score | 56 [49 to 60] | 53 [48 to 58]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were registered at the follow up at 6 months for all participants.
Arm/Group | Iron Isomaltoside 1000 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 1/50
Serious Adverse Events (participants affected / at risk) | 5/52 | 12/50
Other Adverse Events (participants affected / at risk) | 22/52 | 18/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside 1000 (N=52) | Placebo (N=50)
Infection (Infections and infestations) | 0 (0) | 8 (8)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cholelitiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
ST-elevation myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyperthyreosis (Endocrine disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Deceased (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside 1000 (N=52) | Placebo (N=50)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Infection (Infections and infestations) | 12 (12) | 5 (5)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Diabetes (Endocrine disorders) | 1 (1) | 0 (0) — Worsening of diabetes
Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spotty facial discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Syncope (Vascular disorders) | 1 (1) | 0 (0)
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0)
Generalized Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Local rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Left ankle
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Worsening of chronic condition. Did not require hospital admission.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03662789/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT03662789/SAP_001.pdf